CLINICAL TRIAL: NCT00928967
Title: Prospective Multicenter, Non-interventional Study to Evaluate the Impact of the Introduction of Interferon Beta-1 b Treatment on Daily Life Activities in Patients at High Risk of Developing Multiple Sclerosis After a First Clinical Demyelinating Event or Having Received a Confirmed Diagnosis of RRMS
Brief Title: Open, Multicentric, Prospective, Quality of Life Study in Multiple Sclerosis Patients
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 14168; Daily Life Study (Other: company internal); BF0610FR (Other: company internal)
Record Dates: First submitted 2009-06-23; First posted 2009-06-26 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-10

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Quality of life
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1b

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Interferon beta-1b, (Betaseron BAY86-5046)

INTERVENTIONS:
Drug: Interferon beta-1b, (Betaseron BAY86-5046) — The cohort included is described in section 8.5 (inclusion criteria)

SUMMARY:
To evaluate the evolution of the impact on daily life activities over the first 12 months following the introduction of interferon beta-1b treatment in patients presenting RRMS or patients at high risk of developing Multiple Sclerosis after a first clinical demyelinating event

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18 years or over, having received a confirmed diagnosis of RRMS as defined by the MacDonald or Poser criteria or after a first clinical demyelinating event suggestive of Multiple Sclerosis, and meeting the requirements of the study inclusion criteria
* The choice of treatment must be clearly dissociated from the decision to include the patient in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males or females aged 18 years or over, having received a confirmed diagnosis of RRMS as defined by the MacDonald or Poser criteria or after a first clinical demyelinating event suggestive of Multiple Sclerosis, and meeting the requirements of the study inclusion criteria.The choice of treatment must be clearly dissociated from the decision to include the patient in the study.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2007-05; Primary Completion 2010-03 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Evolution of the Daily Life score: Analysis of variance for repeated measurements. | After 1, 3, 6, 9 and 12 months

SECONDARY OUTCOMES:
Evolution of the SF 36 score, Fatigue score, Beck's depression score: analysis of variance for repeated measurements | Over 12 months
Correlation coefficient with quality of life scales | Over 12 months
Kinetics of treatment discontinuation: Kaplan Meier | Over 12 months
Rate of treatment continuation | After 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, France